CLINICAL TRIAL: NCT04313166
Title: A Treatment Continuation Study for Patients With Amyotrophic Lateral Sclerosis/Motor Neuron Disease Who Have Successfully Complete Study CMD-2019-001
Brief Title: Treatment Continuation Study for Patients With ALS/MND Who Completed Study CMD-2019-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD-2020-001
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — copper (II) diacetyl-di(N(4)-methylthiosemicarbazone); Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cu(II)ATSM (Experimental): copper-containing synthetic small molecule
  Interventions: Drug: Cu(II)ATSM

INTERVENTIONS:
Drug: Cu(II)ATSM — cooper-containing synthetic small molecule
  Other Names: diacetylbis(N(4)-methylthiosemicarbazonato) copper(II)

SUMMARY:
Provides up to six months treatment with CuATSM for subjects who have successfully completed study CMD-2019-001

DETAILED DESCRIPTION:
Provides up to six months treatment with CuATSM for subjects who have successffulyl completed study CMD-2019-001. [This allows subjects randomized to placebo on study CMD-2019-001 to receive up to six months treatment with CuATSM and provides an up to an additional six months treatment with CuATSM for subjects randomized to CuATSM on study CMD-2019-001]

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent prior to initiation of any study-specific procedures and treatment
* documented completion of protocol-specified assessments following completion of 24 weeks treatment on study CMD-2019-002
* Investigator considers patient has been tolerating treatment on study CMD-2019-001 and may benefit from continued treatment with CuATSM

Exclusion Criteria:

* not dependent on mechanical ventilation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Treatment-related changes in disease severity | 24 weeks
  Treatment-related changes in disease severity assessed by ALS Functional Rating Scale - Revised (ALSFRS-R)

SECONDARY OUTCOMES:
Treatment-related changes in cognitive function | 24 weeks
  Treatment-related changes in cognitive function by Edinburgh Cognitive and Behavioral Assessment (ECAS) score
Treatment-related changed in respiratory function | SVC
  Treatment-related changes in respiratory function by seated slow vital capacity (SVC)
Treatment tolerance | 24 weeks
  Treatment tolerance based on dose reductions and dose terminations due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Rowe, MD, Principal Investigator — Macquarie University
Locations (1):
- Macquarie University, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No